CLINICAL TRIAL: NCT03183557
Title: Examination of Bone Metabolism and Bone Mineral Density by Zoledronic Acid in Primary and Secondary Osteoporosis
Brief Title: Efficacy of Zoledronic Acid in Osteoporosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shinshu University (Other)
Responsible Party: Principal Investigator, Yukio Nakamura, Associate professor at Shinshu University, Shinshu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Zol2017
Record Dates: First submitted 2017-06-05; First posted 2017-06-12 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Zoledronic Acid; alfacalcidol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ZA alone (Active Comparator)
  Interventions: Drug: "Zoledronic acid", "Reclast®"
- ZA plus VD (Active Comparator)
  Interventions: Drug: "Zoledronic acid", "Reclast®" and "active vitamin D", "alfacalcidol®"

INTERVENTIONS:
Drug: "Zoledronic acid", "Reclast®" — To examine the efficacy of zoledronic acid in osteoporosis
  Arms: ZA alone
Drug: "Zoledronic acid", "Reclast®" and "active vitamin D", "alfacalcidol®" — To examine the efficacy of zoledronic acid plus alfacalcidol in osteoporosis
  Arms: ZA plus VD

SUMMARY:
There has been no comparative data between Zoledronic acid and Zoledronic acid combined with active vitamin D in primary and secondary osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Osteoporotic patients who want to take zoledronic acid

Exclusion Criteria:

* Patients who are allergic to zoledronic acid or vitamin D
* Patients who are pregnant or breast-feeding
* Patients who have not taken zoledronic acid for the last 2 years

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients are separately analyzed
Enrollment: 100 (Estimated)
Dates: Start 2017-10-12 (Actual); Primary Completion 2022-12-08 (Estimated); Study Completion 2025-06-08 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density | Change from Baseline Values at 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Yukio Nakamura, Matsumoto, Nagano, Japan

IPD SHARING:
Plan to Share IPD: No